CLINICAL TRIAL: NCT06862076
Title: The Impact of Lung Function Prehabilitation to Postoperative Pulmonary Complications on Patient Undergoing Upper Abdominal Surgery Treated in Intensive Care Unit: A Randomized Controlled Trial
Brief Title: Impact of Lung Function Prehabilitation to Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Prof. Dr. dr. Dita Aditianingsih, Sp.An-TI., Subsp.T.I.(K)., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IndonesiaUAnes049
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pulmonary Complications (PPCs)
Keywords: Prehabilitation; Postoperative pulmonary complications; Upper abdominal surgery; Intensive care unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Function Prehabilitation (Experimental): Participants assigned to the prehabilitation group received personalized exercise prescriptions, including aerobic training, muscle strengthening, and inspiratory muscle training with a threshold device. The prehabilitation program was conducted at the participants' homes for a minimum duration of two weeks. Adherence was monitored through logbook entries and video call evaluations to ensure correct implementation of the prescribed exercises.
  Interventions: Procedure: Lung Function Prehabilitation
- Standard of Care (No Intervention): No prehabilitation is done, patients in this group received standard of care.

INTERVENTIONS:
Procedure: Lung Function Prehabilitation — Participants assigned to the prehabilitation group received personalized exercise prescriptions, including aerobic training, muscle strengthening, and inspiratory muscle training with a threshold device. The prehabilitation program was conducted at the participants' homes for a minimum duration of two weeks. Adherence was monitored through logbook entries and video call evaluations to ensure correct implementation of the prescribed exercises.
  Arms: Lung Function Prehabilitation

SUMMARY:
The aim of this study is to compare the effect of lung function prehabilitation to postoperative pulmonary complications on patient undergoing upper abdominal surgery treated in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years or older
* scheduled for the upper abdominal surgery under general anesthesia with intraoperative mechanical ventilation
* possess adequate cognitive function to comprehend and follow instructions
* possess sufficient physical capacity to perform structured prehabilitation exercises
* express willingness to participate in the intervention program before surgery

Exclusion Criteria:

* pregnancy
* pre-existing severe pulmonary diseases such as chronic obstructive pulmonary disease (COPD)
* planned laparoscopic procedures
* history of significant neuromuscular impairment (e.g: stroke)
* declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Postoperative day 1 and 3
  Including pulmonary infections, atelectasis, and diaphragmatic dysfunction. Pulmonary infection is assessed using the Clinical Pulmonary Infection Score (CPIS) and with a threshold of >6, atelectasis using Lung Ultrasound Score (LUS) of ≥1, and diaphragm ultrasound were used to evaluate diaphragm ratio. CPIS and LUS score assessments were conducted on postoperative day 1 and 3 by trained investigators, diaphragm ratio assessment was conducted preoperatively and on postoperative day 1 and 3, all findings were systematically recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No